CLINICAL TRIAL: NCT07191964
Title: Assessment of Supra-Sartorial Subcutaneous Infiltration (SSSI) Efficacy When Combined With Intermittent Adductor Canal Block (iACB) and Posterior Capsule Local Infiltration Analgesia (PC-LIA) in Multimodal Pain Management for Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: SSSI Efficacy With iACB and PC-LIA in TKA Pain Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202503094
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain Management in Total Knee Arthroplasty; Peripheral Nerve Blocks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSSI + iACB + PC-LIA (all active) (Active Comparator)
  Interventions: Procedure: Supra-Sartorial Subcutaneous Infiltration (SSSI); Procedure: intermittent adductor canal block (iACB); Procedure: posterior capsule local infiltration analgesia (PC-LIA)
- SSSI (sham) + iACB + PC-LIA (Placebo Comparator)
  Interventions: Procedure: Supra-Sartorial Subcutaneous Infiltration (SSSI); Procedure: intermittent adductor canal block (iACB); Procedure: posterior capsule local infiltration analgesia (PC-LIA)

INTERVENTIONS:
Procedure: Supra-Sartorial Subcutaneous Infiltration (SSSI) — 20 mL ropivacaine or saline infiltrated lateral-to-medial subcutaneously above sartorius at femoral triangle apex using inject-as-you-advance technique, avoiding hyperechoic nerves.
Procedure: intermittent adductor canal block (iACB) — An adductor canal catheter is inserted proximal-to-distally over a distance of 6-10 cm at femoral triangle apex, with an initial bolus of 10 mL of 0.3% ropivacaine administered in PACU. The following doses start at 9:00 PM on the day of surgery and are repeated every 12 hours,
Procedure: posterior capsule local infiltration analgesia (PC-LIA) — PC-LIA consists of two 10 mL injections of 0.3% ropivacaine delivered intraoperatively to the posteromedial and posterolateral aspects of the posterior capsule before cementation. The target injection plane is the potential space between the posterior capsule and the popliteal artery.

SUMMARY:
This prospective, triple-blinded, sham-controlled randomized trial evaluates the additive effect of Supra-Sartorial Subcutaneous Infiltration (SSSI) combined with intermittent adductor canal block (iACB) and posterior capsule local infiltration analgesia (PC-LIA) for pain management in total knee arthroplasty (TKA). SSSI, a simpler alternative to targeted anterior femoral cutaneous nerve (AFCN) block, is tested in 90 adults (45-90 years) randomized into two arms: sham SSSI + active iACB + PC-LIA versus all active interventions. Primary outcome is pain scores on postoperative day 0; secondary outcomes include daily pain trajectory, opioid use, functional recovery, and complications over days 0-3.

DETAILED DESCRIPTION:
This prospective, two-armed, triple-blinded, sham-controlled randomized controlled trial investigates the additive effect of Supra-Sartorial Subcutaneous Infiltration (SSSI) to intermittent adductor canal block (iACB) and posterior capsule local infiltration analgesia (PC-LIA) in multimodal pain management for total knee arthroplasty (TKA). SSSI is a peripheral nerve block technique the investigators devised as a simpler alternative to targeted anterior femoral cutaneous nerve (AFCN) block, which is technically more demanding and time-consuming. Based on the investigators' preliminary study (in publication) where SSSI combined with PC-LIA provided clinically meaningful analgesia in ~58% of patients, and drawing from previous studies on AFCN blocks, the trial compares: Arm 1 (all active SSSI + active iACB + active PC-LIA) versus Arm 2 (sham SSSI + active iACB + active PC-LIA). Adults (45-90 years) undergoing unilateral primary TKA (n=90, 45/arm) will be randomized 1:1, stratified by age, preoperative pain levels (in Numerical Rating Scale) and functional status (WOMAC Index or Knee Society Score). Interventions use 0.3% ropivacaine or saline shams, with SSSI and ACB catheterization performed in the post-anesthesia care unit by anesthesiologists and PC-LIA performed intraoperatively by surgeons. Primary outcome: Numerical Rating Scale pain scores at rest and during continuous passive motion at 9:00 PM on postoperative day (POD) 0, focusing on anteromedial knee pain. Secondary outcomes include daily pain scores, rescue ACB doses, additional opioid use, functional recovery (quadriceps strength, timed up and go [TUG] test), and complications over POD 0-3. With ~96% power for a 2-point NRS difference, this trial evaluates SSSI's role in enhancing motor-sparing analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45-90 undergoing unilateral primary TKA for osteoarthritis.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Able to provide informed consent and use NRS pain scales.
* Surgery scheduled to start before noon to standardize spinal anesthesia recovery.

Exclusion Criteria:

* Bilateral or revision TKA.
* Contraindications to regional anesthesia (e.g., coagulopathy, infection at injection site).
* Chronic opioid use (>30 mg morphine equivalents/day) or preoperative NRS >4.
* Pre-existing neurological deficits in lower extremities or AFCN-related neuropathy.
* Allergy to ropivacaine.
* Pregnancy, breastfeeding, or cognitive impairment affecting assessments.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pain: NRS at rest/movement on postoperative day 0 (with a focus on the anteromedial aspect of knee) | at 9:00 PM on postoperative day 0
  NRS pain scores (0-10) at rest and during continuous passive motion will be taken on postoperative day 0 at 9:00 PM. Higher NRS pain scores indicate worse pain levels.

SECONDARY OUTCOMES:
Pain: NRS at rest/movement (anteromedial vs posterior aspect of knee) from postoperative day 1-3 | From postoperative day 1 at 9:00 AM to postoperative day 3 at 9:00 AM.
  NRS pain scores (0-10) will be taken at rest/during TUG test on postoperative day 1 (9:00 AM, 9 :00 PM), POD 2 (9:00 AM, 9 :00 PM), and POD 3 (9:00 AM). Higher NRS pain scores indicate worse pain levels.
Rescue ACB doses (0.3% ropivacaine, mg) | From the time entering post-anesthesia care unit to postoperative day 3 at 9:00 AM
  Rescue ACB will be administered via catheter as needed outside of the scheduled doses (from postoperative day 0 at 9:00PM to postoperative day 3 at 9:00 AM, q12 hours).
Additional morphine doses (mg) | From the time entering post-anesthesia care unit to postoperative day 3 at 9:00 AM
  Intravenous morphine as bolus or patient-controlled analgesia may be administered as needed if regional anesthesia fails to providing adequate analgesia (NRS pain <4).
Functional: Quadriceps strength (dynamometer), TUG test | From postoperative day 1 at 9:00 AM to postoperative day 3 at 9:00 AM.
  Quadriceps strength will be tested using a dynamometer together with TUG test from postoperative day 1 at 9:00 AM to postoperative day 3 at 9:00 AM, q24 hours
Complications | From postoperative day 0 at 9:00 PM to postoperative day 3 at 9:00 AM.
  Complications such as falls, hematoma/oozing/infection at the catheterization site, catheter dislodgement, etc., will be recorded from postoperative day 0 to postoperative day 3.

OTHER OUTCOMES:
Patient satisfaction | At postoperative day 3 at 9:00 AM.
  Quality of Recovery-15 (QoE-15) scores will be taken on postoperative day 3 at 9:00 AM. Value range 0-150, with the higher scores indicating better recovery.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kampitak W, Tanavalee A, Tansatit T, Ngarmukos S, Songborassamee N, Vichainarong C. The analgesic efficacy of anterior femoral cutaneous nerve block in combination with femoral triangle block in total knee arthroplasty: a randomized controlled trial. Korean J Anesthesiol. 2021 Dec;74(6):496-505. doi: 10.4097/kja.21120. Epub 2021 Jun 29. PMID 34182749
- [Background] Pivec C, Bodner G, Mayer JA, Brugger PC, Paraszti I, Moser V, Traxler H, Riegler G. Novel Demonstration of the Anterior Femoral Cutaneous Nerves using Ultrasound. Ultraschall Med. 2018 Feb 7. doi: 10.1055/s-0043-121628. Online ahead of print. PMID 29415312
- [Background] Bjorn S, Nielsen TD, Jensen AE, Jessen C, Kolsen-Petersen JA, Moriggl B, Hoermann R, Bendtsen TF. The Anterior Branch of the Medial Femoral Cutaneous Nerve Innervates Cutaneous and Deep Surgical Incisions in Total Knee Arthroplasty. J Clin Med. 2024 May 31;13(11):3270. doi: 10.3390/jcm13113270. PMID 38892981
- [Background] Bjorn S, Nielsen TD, Jensen AE, Jessen C, Kolsen-Petersen JA, Moriggl B, Hoermann R, Nyengaard JR, Bendtsen TF. The anterior branch of the medial femoral cutaneous nerve innervates the anterior knee: a randomized volunteer trial. Minerva Anestesiol. 2023 Jul-Aug;89(7-8):643-652. doi: 10.23736/S0375-9393.22.16910-5. Epub 2023 Feb 27. PMID 36852567
- [Background] Bjorn S, Nielsen TD, Moriggl B, Hoermann R, Bendtsen TF. Anesthesia of the anterior femoral cutaneous nerves for total knee arthroplasty incision: randomized volunteer trial. Reg Anesth Pain Med. 2019 Dec 10:rapm-2019-100904. doi: 10.1136/rapm-2019-100904. Online ahead of print. PMID 31826920